CLINICAL TRIAL: NCT04119076
Title: The Effect of a Curriculum-based Physical Activity Intervention on Accelerometer-assessed Physical Activity in Schoolchildren: a Non-randomised Mixed Methods Controlled Before-and-after Study
Brief Title: The Effect of a Curriculum-based Physical Activity Intervention on Physical Activity in Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Alison Innerd, Principal Investigator, Teesside University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TU2019
Record Dates: First submitted 2019-08-21; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Physical Activity
Keywords: school-based intervention; active classroom
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two school allocated to receive the intervention, three schools allocated to the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Teacher delivered a 10 minute classroom-based physical activity on school days for eight weeks.
  Interventions: Other: Classroom-based physical activity
- Control Group (Other): Children in the control schools continued with their usual school routine
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Classroom-based physical activity
  Arms: Intervention Group
Other: Control Group
  Arms: Control Group

SUMMARY:
A non-randomised mixed methods controlled before-and-after study. The study evaluated the effects of a classroom-based physical activity intervention in primary school children on physical activity. Two schools were allocated to deliver the classroom-based intervention for eight weeks, and three schools continued with their usual school routine.

DETAILED DESCRIPTION:
The primary aim of this study was to test the feasibility and potential effect of a classroom-based, curriculum-embedded intervention - ExCiTE; Exercise Classes in the Teaching Environment- on total physical activity and moderate to vigorous physical activity. The secondary aim was to measure and describe health-related quality of life and physical fitness components, and to gain understanding of the experiences, views and attitudes towards the ExCiTE intervention among participating children and schoolteachers.

ELIGIBILITY:
Inclusion Criteria:

* Parental Consent
* Child Assent

Exclusion Criteria:

* Respiratory infections; or.

  * Condition of injury affecting child's ability to undertake exercise
  * Allergic to sticky tape

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Amount of time spent in moderate to vigorous physical activity (MVPA) | Accelerometer (ActiGraph GT3X) worn for 7 days. Analysed using Evenson cutpoints.
  Daily moderate to vigorous physical activity (minutes) collected by wearing an accelerometer for 7 consecutive days.
Total physical activity | Accelerometer (ActiGraph GT3X) worn on the hip for 7 consecutive days. Analysed using Evenson cutpoints
  Total physical activity measured by counts per minute

SECONDARY OUTCOMES:
Aerobic Fitness | 1 Day of testing
  Aerobic Endurance. Multistage fitness test
Health-Related Quality of Life | Recall questionnaire. Questionnaire completed on one day of testing
  27 -item KIDSCREEN questionnaire. Assesses health-related quality of life across five dimensions: physical well-being, psychological well-being, parent relations and autonomy, social support and peers and school environment. Likert Scale 1-5. Test completed at baseline, post-intervention and 4 weeks follow up

OTHER OUTCOMES:
Fitness Test:Balance | Balance for 30 seconds on each leg. Test completed on one day of testing. Participants balances on one leg on a beam for 30 seconds. The number of times the participants has to put the foot on the floor during the 30 seconds is the score.
  Flamingo balance test (from Eurofit Protocol). Stand on a wooden beam for 30 seconds and try to balance for 30 seconds. Complete with each foot
Fitness Test:Flexibility | Best of three attempts on one day of testing.
  Sit and reach test. Sit against the sit and reach box, lean forwards and stretch as far forward as possible. Measured to the nearest cm. The higher the number, the better the flexbility.
Fitness Test: Speed Fitness Test: Speed | one attempt on one day of testing.
  10 x 5m shuttle run (from Eurofit Protocol). Run between two cones 5m apart 10 times. The lower the score, the better
Fitness Test: Hand Eye Coordination | Best of three attempts, one one day of testing. Time is recorded. The faster the time the better the hand eye coordination
  Plate tapping - tap the hand on two different colour spots - using the dominant hand.
Fitness Test: Explosive Strength | Best of three attempts, one one day of testing. Distance is recorded. The further the distance the better the explosive strength
  Standing broad jump. Jump as far forwards as possible keeping both feet together. The measurement is taken from the heel on the furthest back landing foot
Fitness Test: muscular strength and endurance | One day of testing. The number of sit ups completed in 30 seconds. The higher the number equates to a better performance
  Sit up on a mat (from Eurofit Protocol)

IPD SHARING:
Plan to Share IPD: No